CLINICAL TRIAL: NCT02769572
Title: The Effectiveness of Moxibustion Treatment for Osteoarthritis of the Knee : a Double-blinded, Double-dummy, Randomized Controlled Trial
Brief Title: Moxibustion in Osteoarthritis of the Knee
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chengdu University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015CB55450401
Record Dates: First submitted 2016-05-10; First posted 2016-05-11 (Estimated); Last update posted 2020-02-17 (Actual); Status verified 2020-02

CONDITIONS: Knee Osteoarthritis
Keywords: Knee osteoarthritis; moxibustion; diclofenac sodium gel
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- real moxibustion plus placebo gel (Experimental): In subjects with osteoarthritis of the knee
  Interventions: Other: real moxibustion; Drug: placebo gel
- diclofenac sodium gel plus sham moxibustion (Active Comparator): In subjects with osteoarthritis of the knee
  Interventions: Drug: diclofenac sodium gel; Other: sham moxibustion

INTERVENTIONS:
Other: real moxibustion — 3 times a week for 4 consecutive weeks,totally 12 sessions at 3 acupoints (ST35, EX-LE4, ST36 )
  Arms: real moxibustion plus placebo gel
Drug: placebo gel — 4 grams per knee, 4 times per day, for 4 weeks
  Arms: real moxibustion plus placebo gel
Drug: diclofenac sodium gel — 4 grams per knee, 4 times per day, for 4 weeks
  Arms: diclofenac sodium gel plus sham moxibustion
Other: sham moxibustion — 3 times a week for 4 consecutive weeks,totally 12 sessions at 3 acupoints (ST35, EX-LE4, ST36 )
  Arms: diclofenac sodium gel plus sham moxibustion

SUMMARY:
This is a multicenter , double-blinded, double-dummy, randomized controlled clinical trial to evaluate the efficacy of moxibustion for osteoarthritis of the knee.

DETAILED DESCRIPTION:
Aim: To evaluate the effectiveness of moxibustion treatment for patients with osteoarthritis of the knee, with respect to relieving pain, improving the dysfunction and improving their quality of life as well.

Design: A multicentre, double-blinded, double-dummy, randomized controlled clinical study will be performed in China. Eligible participants will be randomly assigned to moxibustion group (real moxibustion plus placebo gel) and the control group (diclofenac sodium gel plus sham moxibustion) with a 1:1 allocation ratio. Participants in both groups will receive 12 sessions of real/sham moxibustion in 4 weeks at 3 acupoints (ST35, EX-LE4, ST36 ). Either diclofenac sodium gel or placebo gel will be applied 4 g per knee 4 times daily for 4 weeks. The whole study period is 13 weeks, with a 1-week run-in period, 4-week treatment phase, and 8-week follow-up phase. The primary outcome measure will be the change of the global scale of the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) at the end of the course. The secondary outcomes include the change of other subscales (pain, stiffness, and function) of WOMAC, Visual Analogue scale (VAS) and Patient Global Assessment (PGA). Safety will be assessed at every visit.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged between 40 and 75 years, with knee osteoarthritis diagnosed according to American College of Rheumatology criteria
* Radiologic confirmation of osteoarthritis in 1 or both knees (Kellgren-Lawrence score 2 or 3)
* Had knee pain in one or both knee(s) of longer than 3 months'duration
* The average severity of knee pain at least 3 points on a10-point of visual analogue scale(VAS)
* Never experienced moxibustion before this trial
* Participants who are willing to comply with our study protocol
* Participants who agree to sign the consent form

Exclusion Criteria:

* Subjects with serious diseases including cancer, uncontrolled hypertension, diabetes mellitus requiring insulin injection, life-threatening cardiovascular or neurological events, chronic respiratory disease, a haemorrhagic disorder and serious mental diseases
* Subjects had pain in the knee may caused by inflammatory, malignant, autoimmune disease or traumatic injury;
* Subjects received knee replacement surgery for the affected knee
* Subjects received knee arthroscopy within the past year, steroid or hyaluronic acid injection in the knee joints within the previous 3 months
* Subject who currently participate in another clinical trial
* Subjects received physiotherapy or other treatments for osteoarthritis knee pain (with the exception of non-steroidal anti-inflammatory drugs) during the previous 4 weeks;

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
The change of the global scale of the Western Ontario and McMaster Osteoarthritis Index (WOMAC) | 4 weeks from baseline

SECONDARY OUTCOMES:
The changes from baseline to 2, 4, 8,12 weeks in the WOMAC subscales (pain, stiffness, and function) | at baseline(0 week), 2 weeks, 4weeks, 8 weeks and 12 weeks later after allocation
The change from baseline to 2, 4, 8,12 weeks in Visual Analogue Scale for the pain intensity. | at baseline(0 week), 2 weeks, 4weeks, 8 weeks and 12 weeks later after allocation
The change of Patient global assessment score | 2 weeks, 4weeks, 8 weeks and 12 weeks later after allocation

CONTACTS AND LOCATIONS:
Overall Officials: Yong Tang, Professor, Study Director — Chengdu University of Chinese Traditional Medicine; Jianying Zhou, Principal Investigator — Chengdu University of Chinese Traditional Medicine
Locations (1):
- Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Zhou JY, Luo L, Zhu LL, Yin HY, Wu Q, Peng JX, Zhang CS, Lv P, Tang Y, Yu SG. Moxibustion versus diclofenac sodium gel for the treatment of knee osteoarthritis: a study protocol for a double-blinded, double-placebo, randomised controlled trial. BMJ Open. 2017 Apr 12;7(4):e012879. doi: 10.1136/bmjopen-2016-012879. PMID 28404609